CLINICAL TRIAL: NCT06193135
Title: Usefulness of Corifollitropin α as Alternative to Conventional Daily rFSH Protocols in Oocyte Donors Undergoing Pituitary Suppression With Medroxiprogesterona Acetate (MPA)
Acronym: TROPIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2304-VLC-051-JG
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Infertility, Female; Reproductive Sterility
Keywords: Oocyte donation; Corifolitropin alpha; Premature luteinization; Medroxiprogesterone acetate; Controlled ovarian estimulation; Folitropin beta
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — follitropin beta

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, open-label, parallel-group, low-intervention, single-center clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elonva (Experimental): Patients will undergo controlled ovarian stimulation with Corifolitropin α (Elonva), 100-150 micrograms (100 in< 60kg and 150 ≥ 60 kg) + Progevera 10 mg.
  Interventions: Drug: Corifolitropin Alfa
- Puregon (Active Comparator): Patients will undergo controlled ovarian stimulation with Folitropin β (Puregon) + Progevera 10 mg.
  Interventions: Drug: Folitropin Beta

INTERVENTIONS:
Drug: Corifolitropin Alfa — Patients will receive a single dose of Colifolitropin alfa, then will receive daily dose of Folitropin Beta since triggering criteria are met.
  Other Names: ELONVA
  Arms: Elonva
Drug: Folitropin Beta — Patient will receive daily dose of Folitropin Beta since triggering criteria are met.
  Other Names: PUREGON
  Arms: Puregon

SUMMARY:
IVF patients frequently experience physical, emotional or physicological burden; this is particularly relevant in the case of oocyte donors, since young women undergo a procedure that is of no health benefit to them. One of the phases of the treatment that contributes most to this situation is ovarian stimulation; as it involves the administration of daily injections which, in addition to the discomfort of administration, causes anxiety to the patient about its correct administration and possible side effects and to physicians concerns about patient compliance.

Advances in pharmacology and knowledge of ovarian pathophysiology have led to the development of new protocols that simplify and reduce drug administration, decrease the potential risk of misapplication and contribute to an improved patient experience. In this context, Corifollitropin α, a long-acting recombinant FSH (rFSH) molecule, provides with a single subcutaneous injection similar results as daily administration of rFSH during a week.

On the other hand, conventional stimulation protocols used in ART resort to using a GnRH analogue (agonist or antagonist) to prevent early luteinization, which is defined as the presence of a progesterone value of > 1.5 ng/ml on the day of induced ovulation. Nevertheless, its use presents some disadvantages, such as it being sometimes complex to achieve desensitization or consistent hypothalamic block, risk of OHS when ovulation is triggered with HCG or its cost. Hence the interest in exploring new options to prevent a premature peak in LH. Nowadays, the oral administration of progestagens (progesterone-primed ovarian stimulation [PPOS]) during the follicular phase of ovarian stimulation (OS) has emerged as an attractive alternative to conventional protocols for preventing early luteinization. Moreover, PPOS produces a similar or even better, in some subgroups, response to OS (length of treatment, number of MII, cancelation rate, etc.), reproductive outcomes (pregnancy rate, live birth rate, etc) and safety (rate of ovarian hyperstimulation [OHSS] or congenital malformations).

Thus, PPOS would seem to be an effective option for personalized protocols, particularly when fresh embryo transfer (FET) is not to be performed, a circumstance that is likely to rise in frequency given the progressive increase in women's age at childbearing; for example, in oocyte donation, or in fertility preservation (FP) and preimplantation genetic testing for aneuploidy (PGT-A). However, very little data are available regarding cycle outcome following Corifollitropin α and PPOS as pituitary suppressor.

The present study, a prospective RCT, was designed to evaluate cycle characteristics (MII oocytes as the primary objective) and endocrinologic profiles of oocyte donors receiving Corifollitropin α and MPA as co-treatment compared with those receiving a daily dose of rFSH (follitropin β) as a control.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the subject's informed consent prior to any trial-related activity.
* Age between 18 and 35 years (both inclusive).
* Regular menstrual cycle, from 25 to 35 days (both inclusive).
* Absence of physical and psychological illness at the time of donation at the discretion of the investigator.
* BMI 18-28 kg/m2 (both inclusive) at the time of donation.
* No personal or family history of interest at the discretion of the investigator.
* Normal uterus and ovaries, without organic pathology.
* No polycystic ovaries.
* Antral follicle count greater than 12 in the sum of the two ovaries at the time of the screening visit.
* Normal karyotype.
* Negative infectious disease screening (Hepatitis B Virus, Hepatitis C Virus, Human Immunodeficiency Virus and Syphilis).
* General analysis with hemogram, hemostasis and biochemistry with parameters within normality.

Exclusion Criteria:

* Concurrent participation in another clinical trial.
* Previous participation in this clinical trial.
* Use of long-term hormonal contraception (hormonal IUD or subcutaneous implants) at least 1 month prior to enrollment.
* Any systemic or metabolic disorder (i.e.: diabetes...) that contraindicates the use of gonadotropins.
* Personal history of thrombophlebitis and thromboembolic phenomena and hypertension.
* Severe hepatic insufficiency, cardiovascular disease
* Suspicion or evidence of breast malignancy or hormone-dependent genital organs.
* Known hypersensitivity to AMP or its excipients
* Any reason for exclusion from the oocyte donation program.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the number of total oocytes obtained after controlled ovarian stimulation with α-Corifolitropin vs. β-Folitropin in donors in whom medroxyprogesterone acetate (MPA) was used to prevent early luteinization. | 2 years
  Number of total oocytes and oocytes metaphase II
To compare the number of metaphase II (MII) oocytes obtained after controlled ovarian stimulation with α-Corifolitropin vs. β-Folitropin in donors in whom medroxyprogesterone acetate (MPA) was used to prevent early luteinization. | 2 years
  Quantification of total oocytes in metaphase II

SECONDARY OUTCOMES:
Incidence of early luteinization | 2 years
  Quantification of cycle cancellation due to lack of response and failure to obtain MII oocytes in puncture.
Medication tolerance: pain, abdominal distension, ovarian hyperstimulation syndrome (OHSS), etc. | 2 years
  Quantification of pain, abdominal distension, ovarian hyperstimulation syndrome (OHSS) using a specifically designed questionarie for this strudy.
Controlled ovraian stimulation duration | 2 years
  Quantification of total days of estimulation
Total cost of each stimulation type. | 2 years
  Quantification of cost.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - IVI Valencia, Valencia, Valencia
  - Ivi Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalfoglou AL. Navigating conflict of interest in oocyte donation. Am J Bioeth. 2001 Fall;1(4):W1. doi: 10.1162/152651601317139333. No abstract available. PMID 12858870
- [Background] Requena A, Cruz M, Collado D, Izquierdo A, Ballesteros A, Munoz M, Garcia-Velasco JA. Evaluation of the degree of satisfaction in oocyte donors using sustained-release FSH corifollitropin alpha. Reprod Biomed Online. 2013 Mar;26(3):253-9. doi: 10.1016/j.rbmo.2012.11.015. Epub 2012 Dec 5. PMID 23352098
- [Background] Corifollitropin alfa Ensure Study Group. Corifollitropin alfa for ovarian stimulation in IVF: a randomized trial in lower-body-weight women. Reprod Biomed Online. 2010 Jul;21(1):66-76. doi: 10.1016/j.rbmo.2010.03.019. Epub 2010 Mar 28. PMID 20483664
- [Background] Boostanfar R, Shapiro B, Levy M, Rosenwaks Z, Witjes H, Stegmann BJ, Elbers J, Gordon K, Mannaerts B; Pursue investigators. Large, comparative, randomized double-blind trial confirming noninferiority of pregnancy rates for corifollitropin alfa compared with recombinant follicle-stimulating hormone in a gonadotropin-releasing hormone antagonist controlled ovarian stimulation protocol in older patients undergoing in vitro fertilization. Fertil Steril. 2015 Jul;104(1):94-103.e1. doi: 10.1016/j.fertnstert.2015.04.018. Epub 2015 May 21. PMID 26003273